CLINICAL TRIAL: NCT01018550
Title: A Randomized, Double-Blind, Placebo Controlled, Multiple Dose Phase 2 Study to Determine the Safety and Efficacy of AMG 853 in Subjects With Inadequately Controlled Asthma
Brief Title: AMG 853 Phase 2 Study in Subjects With Inadequately Controlled Asthma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20080615
Record Dates: First submitted 2009-11-19; First posted 2009-11-23 (Estimated); Last update posted 2016-03-23 (Estimated); Status verified 2016-02

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — vidupiprant

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- AMG 853 (Experimental)
  Interventions: Drug: AMG 853
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AMG 853 — AMG 853 5 mg (BID)
  Arms: AMG 853
Drug: AMG 853 — AMG 853 200 mg (QD)
  Arms: AMG 853
Drug: AMG 853 — AMG 853 25 mg (BID)
  Arms: AMG 853
Drug: AMG 853 — AMG 853 100 mg (BID)
  Arms: AMG 853
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The primary objective is to determine if AMG 853 is effective compared with placebo as measured by change in Asthma Control Questionnaire (ACQ) composite symptoms scores from baseline to week 12.

ELIGIBILITY:
Inclusion Criteria:

* Males or females 18 to 65 years of age
* Percent of predicted FEV1 ≥ 50% and ≤ 80%
* At least 12% reversibility over pre-bronchodilator FEV1
* Inhaled corticosteroid (ICS) ≥ 200 and ≤ 1000 µg/day fluticasone or equivalent.
* Ongoing asthma symptoms with ACQ score ≥ 1.5 points

Exclusion Criteria:

* History of chronic obstructive pulmonary disease or other chronic pulmonary condition other than asthma
* Any uncontrolled, clinically significant systemic disease
* Respiratory infection within 4 weeks of the screening visit

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 397 (Actual)
Dates: Start 2009-10; Primary Completion 2010-12 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
The primary objective is to determine if AMG 853 is effective compared with placebo as measured by change in Asthma Control Questionnaire (ACQ) composite symptoms scores from baseline to week 12. | Baseline to Week 12

SECONDARY OUTCOMES:
Evaluate the efficacy of AMG 853 as measured by use of rescue short-acting β-agonist (SABA) | Baseline to Week 12
Evaluate the efficacy of AMG 853 as measured by daily symptom score (aggregate/night and individual symptoms; and symptom free days) | Baseline to Week 12
Evaluate the efficacy of AMG 853 as measured by pre- and post-bronchodilator forced expiratory volume in 1 second (FEV1) | Baseline to Week 12
Evaluate the efficacy of AMG 853 as measured by AM and PM peak expiratory flow rate (PEFR) | Baseline to Week 12
Evaluate the efficacy of AMG 853 as measured by asthma quality of life questionnaire (AQLQ) | Baseline to Week 12

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Background] Busse WW, Wenzel SE, Meltzer EO, Kerwin EM, Liu MC, Zhang N, Chon Y, Budelsky AL, Lin J, Lin SL. Safety and efficacy of the prostaglandin D2 receptor antagonist AMG 853 in asthmatic patients. J Allergy Clin Immunol. 2013 Feb;131(2):339-45. doi: 10.1016/j.jaci.2012.10.013. Epub 2012 Nov 20. PMID 23174659
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com